CLINICAL TRIAL: NCT06461546
Title: Imlifidase in Living Donor Renal Transplantation Highly Sensitized Recipients (LIVEDES)
Brief Title: Imlifidase in Living Donor Renal Transplantation Highly Sensitized Recipients
Acronym: LIVEDES
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to provide study drug to participants
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIVEDES study; 2024-513607-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplant Candidates
Keywords: living kidney trasplant; imlifidase treatment
MeSH Terms: interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Intervention Model Description: Phase II, prospective, single arm pilot study. To evaluate the ability of Imlifidase treatment to achieve a negative virtual crossmatch in patients with available live donor kidney.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imlifidase treatment (Experimental): Single arm pilot study
  All highly sensitized patients included in the study will receive the immunosuppressive standard of care therapy at Hospital Clínic de Barcelona and in addition the study drug:
  * Imlifidase (POD0, pre-transplantation), imlifidase, 0.25 mg/kg over a period of 15 minutes, prior to transplantation.
  * Dose Adjustment Criteria
  FC-XM screening and single antigen will be performed after 6 hours of imlifidase infusion, It will take 3 hours to obtain the results, respectively:
  * NEGATIVE (FC-XM) - renal transplantation will be performed as soon as possible.
  * POSITIVE (FC-XM) - 2nd Imlifidase infusion will be required (imlifidase dose: 0.25mg/Kg).
  FC-XM screening and single antigen will be performed after 2 hours of the 2nd Imlifidase infusion:
  * NEGATIVE (FC-XM) - renal transplantation will be performed as soon as possible.
  * POSITIVE (FC-XM) - The scheduled kidney transplant will be canceled.
  Interventions: Drug: Imlifidase

INTERVENTIONS:
Drug: Imlifidase — * Imlifidase (POD0, pre-transplantation), imlifidase, 0.25 mg/kg over a period of 15 minutes, prior to transplantation.
  * Dose Adjustment Criteria
  FC-XM screening and single antigen will be performed after 6 hours of imlifidase infusion, It will take 3 hours to obtain the results, respectively:
  * NEGATIVE (FC-XM) - renal transplantation will be performed as soon as possible.
  * POSITIVE (FC-XM) - 2nd Imlifidase infusion will be required (imlifidase dose: 0.25mg/Kg).
  FC-XM screening and single antigen will be performed after 2 hours of the 2nd Imlifidase infusion:
  * NEGATIVE (FC-XM) - renal transplantation will be performed as soon as possible.
  * POSITIVE (FC-XM) - The scheduled kidney transplant will be canceled.

SUMMARY:
This is a Phase II, pilot, prospective, unicentric trial, to evaluate Imlifidase could improve the transplantability of the highly sensitized patients with good outcomes respect to survival and functionality of the graft.

DETAILED DESCRIPTION:
The patients between 18 and 65 years will be flow cytometry crossmatch (FC-XM) positive against an available living donor. The imlifidase treatment will turn the crossmatch test negative prior to transplantation. A second dose of imlifidase can be given within 24 hours if the first dose is considered not to have sufficient effect. If a second dose is given, a confirmatory FCXM test will be performed pre-second imlifidase dosing and between 2-6 hours following the second dose.

ELIGIBILITY:
Inclusion Criteria:Inclusion Criteria To be eligible to participate in this study, candidates must meet the following elegibility criteria. Currently, at the Hospital Clinic of Barcelona, up to 10 highly sensitized patients would meet the following inclusion criteria.

* Participant Inclusion Criteria
* Sensitized (cPRA ≥ 50%) kidney transplant candidates between 18 and 65 years.
* Low probability to get a transplant in a kidney exchange program (KEP) from a living donor.
* Included in the living donor program, with an accepted potential living donor.
* Donor and recipient must meet the eligibility criteria for donation and kidney transplantation respectively at the Hospital Clinic of Barcelona and the national guidelines.
* Presence of donor-specific antibody/crossmatch positive (DSA/FC-XM+) non-HLA identical donor.

  * at least one DSA with MFI >3.000.
  * and DSA MFI <10.000 (in serum samples diluted 1/64).
  * and maximum two Class II DSAs.
  * and maximum 17 points in Jordan RIS Score (DSA 2500-5000: 2 points; DSA MFI 5001-10000: 5 points; DSA MFI > 10000: 10 points)
* Women of childbearing age must take contraceptive measures because Imlifidase is not recommended during pregnancy.
* Must have given written informed consent (signed and dated) and any authorizations required by local law and be able to comply with all study requirements.

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from participation in this study:

• Participant Exclusion Criteria

1. Known contraindications for therapy with IVIG, Rituximab, plasma exchange (PLEX) or Imlifidase.
2. Recipients of Deceased Donors (DBD, Extended Criteria Donors (ECD) or DCD).
3. A positive Complement-Dependent Cytotoxicity (CDC) Crossmatch against the living donor.
4. HIV-positive subjects.
5. Subjects who test positive for HBV infection [positive HBVsAg or HBVeAg/DNA] or HCV infection [RNA+].
6. Subjects with active TB.
7. Subjects with selective IgA deficiency, those who have known anti-IgA antibodies, and those with a history of anaphylaxis or severe systemic responses to any part of the clinical trial material.
8. Subjects who have received or for whom multiple organ transplants are planned.
9. A significantly abnormal general serum screening lab result defined as WBC<3.0x103/ml, Hgb<8.0 g/dL, platelet count <100x103/ml, SGOT>3xupper limit.
10. Subjects with active CMV or EBV infection as defined by positive PCR.
11. Subjects with a known history of previous myocardial infarction within one year of screening.
12. Subjects with a history of clinically significant thrombotic episodes, and subjects with active peripheral vascular disease.
13. Patients with a kidney disease with high risk of recurrence and/or complement-associated kidney disease (aHUS, etc).
14. Subjects with Protein C and Protein S deficiency.
15. Pregnant and lactating women
16. Current diagnosis or history of thrombotic thrombocytopenic purpura (TTP), or known familial history of TTP.
17. Known allergy to Imlifidase or excipient of the drug preparation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
• Proportion of patients with conversion of a positive virtual crossmatch to negative within 6 hours after imlifidase treatment (up to two doses). | 6 hours
  The fraction of patients with a conversion of a positive FC-XM within 6 hours of treatment with imlifidase.

SECONDARY OUTCOMES:
1. Proportion of patients that require a second dose of imlifidase | 24 hours
  To evaluate flow cytometry T-cell crossmatch conversion within 24 hours of imlifidase treatment, requirement of a second dose of imlifidase.
2. To evaluate the rebound of preexisting donor specific antibodies (DSA) (difference between MFI of each DSA daily - until D+14 - compared to pre-imlifidase administration) | daily, from day 0 to day 14
  Pre-existing DSA appearance measured daily until D+14
3. De novo DSA appearance over 14 days after imlifidase treatment | daily, from day 0 to day 14
  To evaluate the appearance of de novo DSAs (any DSA no present in pre-transplant or historical) daily - until D+14. To be considered positive the bead MFI should be over 750 and to be above the bead specific threshold related to the lowest bead of the same locus.
4. To evaluate HLA/DSA antibody levels up to 1 year after transplantation | time points between pre-dose imlifidase and 2 weeks, and at 1, 3 and 6 months and 1 year after imlifidase treatment
  HLA/DSA antibody levels at several time points between pre-dose imlifidase and 2 weeks, and at 1, 3 and 6 months and 1 year after imlifidase treatment
5. To evaluate renal function up to 1 year after transplantation | time points between 24 hours and 2 weeks and at 1, 3 and 6 months and 1 year after transplantation as assessed
  by estimated glomerular filtration rate (eGFR) and serum/plasma creatinine levels
6. To evaluate patient survival 1 year after transplantation | at 12 months after transplantation
  Patient survival at 12 months after transplantation
7. To evaluate the graft survival at 12 months | at 12 months after transplantation
  To evaluate the graft survival at 12 months (both overall and death-censored analysis).
8. Proportion of patients with biopsy confirmed rejection, either cell-mediated or antibody-mediated rejection, over 1 year | within 12 months
  To evaluate the incidence of acute allograft rejection within 12 months (overall and stratified by type: cell mediated rejection or antibody-mediated rejection
9. To evaluate safety of Imlifidase treatment with regards to infusion related reactions occurring within 48 hours of Imlifidase infusion | within 48 hours of Imlifidase infusion
  Proportion of patients with infusion-related reactions within 48 hours of Imlifidase infusion
10.adverse events within 30 days after transplantation | 30 days after transplantation
  Proportion of patients with adverse events within 30 days after transplantation
11. Proportion of patients with severe or serious infections | 6 months and 12 months
  To evaluate the adverse events ( infectious disease that required hospitalization) at 6 and 12 months.
12. To evaluate safety of Imlifidase treatment with regards to reported serious adverse events (SAEs) | 12 months
  Safety over 1 year as measured by reported SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Diekmann, Dr, Principal Investigator — Fundació de Recerca Clínic Barcelona - Institut D'Investigacions Biomèdiques Agustí Pí i Sunyer

IPD SHARING:
Plan to Share IPD: No